CLINICAL TRIAL: NCT01901536
Title: Promotion of Coparenting During Family Formation Period
Brief Title: Family Foundations Coparenting Pilot Trial
Acronym: FF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Mark Feinberg, Research professor, Feinberg, Mark, Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH64125-01A2
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Parent-Child Relations
Keywords: First time parents; Coparenting; Family Foundations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Couples randomly assigned to the Intervention Group received the Family Foundations Coparenting Program.
  Interventions: Behavioral: Family Foundations Coparenting Program
- Control Group (No Intervention): Couples in the Control group did not receive the Family Foundations Coparenting Program.

INTERVENTIONS:
Behavioral: Family Foundations Coparenting Program — Family Foundations, a program for adult couples expecting their first child, is designed to help them establish positive parenting skills and adjust to the physical, social, and emotional challenges of parenthood. Program topics include coping with postpartum depression and stress, creating a caring environment, and developing the child's social and emotional competence.
  Family Foundations is delivered to groups of couples through four prenatal and four postnatal classes of 2 hours each. Prenatal classes are started during the fifth or sixth month of pregnancy, and the postnatal classes end when the children are 6 months old.
  Family Foundations is delivered in a community setting by childbirth educators who have received 3 days of training from Family Foundations staff.
  Arms: Intervention Group

SUMMARY:
This is a research study to evaluate the effectiveness of the Family Foundations program and to better understand how families cope with having a new baby. The research questions include: What is the effectiveness of the Family Foundations program? How do families cope with having a new baby?

ELIGIBILITY:
Inclusion Criteria:

* Expecting first child
* Couple living together and planning to raise child together
* 18 years or older

Exclusion Criteria:

* Not first child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2002-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Coparenting Quality | up to 3.5 years after baseline
  We assessed coparenting relationship quality with the 31-item Coparenting Scale, which was created based on prior work (e.g., Abidin & Brunner, 1995; Cordova, 2001; Frank, Olmstead, Wagner,& Laub, 1991; Margolin et al., 2001; McHale, 1997). The overall score represents an average of items covering theoretically important domains: coparental agreement, support,undermining, and exposure of the child to conflict.

SECONDARY OUTCOMES:
Parenting Discipline Practices | 3.5 years after baseline
  The Parenting Scale assesses discipline practices in parents of children from 18-48 months (Arnold,O'Leary, Wolff, & Acker, 1993).
Child Behavior Problems | 3.5 years after baseline
  Child behavior problems were measured using the Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2000), reported by mothers only. From this 100-item questionnaire, separate sub-scales were calculated using scoring conventions. From these, we examined three overall scores which were normed for child age:
  Total problems, Externalizing problems, and Internalizing problems. In addition, we examined two specific sub-scales given their relevance to this study: Aggression and Attention/Hyperactivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, Prevention Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Result] Feinberg ME, Jones DE, Kan ML, Goslin MC. Effects of family foundations on parents and children: 3.5 years after baseline. J Fam Psychol. 2010 Oct;24(5):532-42. doi: 10.1037/a0020837. PMID 20954763
- [Result] Feinberg ME, Kan ML, Goslin MC. Enhancing coparenting, parenting, and child self-regulation: effects of family foundations 1 year after birth. Prev Sci. 2009 Sep;10(3):276-85. doi: 10.1007/s11121-009-0130-4. PMID 19381809
- [Result] Feinberg ME, Kan ML. Establishing family foundations: intervention effects on coparenting, parent/infant well-being, and parent-child relations. J Fam Psychol. 2008 Apr;22(2):253-63. doi: 10.1037/0893-3200.22.2.253. PMID 18410212
- [Derived] Moran LJ, Lee JK, Jones D, Fronberg K, Feinberg ME. Coparenting-focused preventive intervention reduces postnatal maternal BMI and buffers impact of cortisol. Obesity (Silver Spring). 2022 Aug;30(8):1564-1572. doi: 10.1002/oby.23466. Epub 2022 Jul 19. PMID 35854331
- [Derived] Roettger ME, Schreier HMC, Feinberg ME, Jones DE. Prospective Relations Between Prenatal Maternal Cortisol and Child Health Outcomes. Psychosom Med. 2019 Jul/Aug;81(6):557-565. doi: 10.1097/PSY.0000000000000705. PMID 31058707